CLINICAL TRIAL: NCT00646022
Title: Natural History of Familial Carcinoid Tumor
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080098; 08-DK-0098
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-21

CONDITIONS: Carcinoid
Keywords: Neuroendocrine; PET; Gastrointestinal; Serotonin; Natural History; Carcinoid Tumor; Gastrointestinal Carcinoid Tumor; Familial Cancer Tumor
MeSH Terms: conditions — Carcinoid Tumor | interventions — fluorodopa F 18

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Participants who undergo extended evaluation for disease at NIH
  Interventions: Drug: [18F]-DOPA
- Arm 2: Participants who do not undergo extended screening or evaluation for disease at NIH
  Interventions: Drug: [18F]-DOPA

INTERVENTIONS:
Drug: [18F]-DOPA — 18F-DOPA PET/CT Scan.

SUMMARY:
This study will evaluate members in families with a history of small bowel carcinoid cancer to study the natural history of those family members that have the disease, determine ways to improve early detection by performing surveillance on those at risk but without disease and to identify the gene(s) that may cause the tumors. Familial carcinoid tumors usually originate in hormone-producing cells that line the small intestine or other cells of the digestive tract. The tumors are slow-growing and usually take many years before they cause symptoms. It is known that these tumors occur more often in some families and are then passed from one generation to the next by inherited genes.

Members of families, including all siblings and offspring in which two or more immediate blood relatives have had small bowel carcinoid tumors are eligible for this study. In some cases unaffected spouses of family members diagnosed with carcinoid cancer are also requested to participate by donating a sample of blood only.

Participants undergo a medical evaluation every 3 years during a 3- to 5-day hospital stay at the NIH Clinical Center. All participants have a personal and family medical history obtained and undergo a physical examination, blood and urine tests.

People who already have a small bowel carcinoid tumor or are at risk of developing a carcinoid tumor have some or all of the following procedures to determine the presence of carcinoid tumor and its (omit next two words- location or) spread to other areas of the body:

* Video Capsule Endoscopy: Visualization of the gastrointestinal tract by ingesting a disposable, "vitamin-pill sized" video capsule that has its own camera and light source.
* CT of the chest abdomen and pelvis with oral and IV contrast : X-ray examination of the chest, abdominal and pelvis organs.
* 18 FDOPA Positron emission tomography (PET) with CT for localization: Nuclear imaging scan to look at tumor activity.
* MRI Liver with contrast - to determine if disease has spread to liver
* Gallium 68 PET/CT-limited to individuals that have residual tumor.
* Clinical and research blood work

Should mid gut carcinoid tumors be found every participant will be assisted in determine what the best course of treatment will be for them.

DETAILED DESCRIPTION:
Study Description:

This study is designed as a prospective evaluation for diagnostic screening, genotyping and natural history of participants belonging to kindreds with familial carcinoid tumor.

Objectives:

Primary Objective:

Study the natural history of familial carcinoid tumors: incidence, age of onset, symptoms, the appropriate diagnostic (biochemical and imaging) modalities, location, histology and metastatic potential of the tumors, metabolic sequelae of the tumor, and clinical and biochemical prognostic factors.

Secondary Objectives:

* Screen for occult disease and determine whether early detection affects the natural history of the disease.
* Compare the sensitivity and specificity of various imaging tomography (CT) with IV contrast and oral Breeza, 18F-DOPA PET/CT scan, [68Ga] DOTATATE PET/CT scan and endoscopic modalities for diagnosing and following carcinoid tumors.
* Collect tumor specimens for histologic evaluation, culturing of intestinal organoids, and genotyping (including DNA and RNA sequencing).
* Sequester DNA from peripheral blood for genotyping (including sequencing) with the intention of localizing a susceptibility gene/s responsible for the familial occurrence of the disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

There are four types of participants who will be included in this protocol as outlined below.

In order to be eligible to participate in this study, an individual must meet all of the following criteria for their group:

Group 1 (Arm 1 or Arm 2)

* Male and female subjects >= 18 years of age
* Have a diagnosis of small intestinal carcinoid tumor
* Have at least one blood relation with a diagnosis of either small intestinal, pulmonary, kidney or gastropancreatic neuroendocrine tumor or metastatic neuroendocrine tumor of unknown primary

Group 2 (Arm 1 or Arm 2)

* Male and female subjects >= 18 years of age
* Has multiple synchronous primary small intestinal tumors

Group 3 (Arm 1 or Arm 2)

* Male and female subjects >=18 years of age
* Does not have a diagnosis of carcinoid tumor
* Has one of the following:

  * at least two blood relatives with any combination of diagnoses of small intestinal carcinoid tumor, a pulmonary, kidney, gastropancreatic neuroendocrine tumor or metastatic neuroendocrine tumor of unknown primary OR
  * has at least one blood relative with multiple, synchronous primary small bowel tumors

Group 4 (Arm 2 only)

* Male and female subjects >= 18 years of age
* Not biologically related to the participating family but has offspring who is/are blood relative(s) of a participating subject.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

1. Members of families with multiple endocrine neoplasia (MEN) I, MEN II or other familial tumor syndromes such as Von Hippel Lindau Syndrome and Neurofibromatosis type I and type II for which there is a known genetic predisposition to non-carcinoid tumors as well as

   carcinoid tumors will be excluded from the study.
2. Any condition which, in the opinion of the investigator, would make it unsafe to participate or would prohibit completion of the protocol.
3. Inability to provide informed consent (Arm 1 only)
4. Pregnant or breastfeeding (Arm 1 only)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2008-08-25 (Actual)

PRIMARY OUTCOMES:
Study the natural history of familial carcinoid tumors | End of study
  Incidence, age of onset, symptoms, the appropriate diagnostic (biochemical and imaging) modalities, location, histology and metastatic potential of the tumors, metabolic sequelae of the tumor, and clinical and biochemical prognostic factors

SECONDARY OUTCOMES:
Compare the sensitivity and specificity of various imaging modalities: computed tomography (CT) with IV contrast and oral Volumen, 18F-DOPA PET/CT scan, [68Ga]DOTATATE PET/CT scan and endoscopic modalities for diagnosing and following carcinoid ... | End of study
  Enrollment of a sufficient number of subjects to allow for the determination of sensitivity and specificity for each imaging and endoscopic modality to show statistically significant superiority for one modality relative to the others
Sequester DNA from peripheral blood for genotyping (including sequencing) with the intention of localizing a susceptibility gene/s responsible for the familial occurrence of the disease | End of study
  Determination of the gene mutation responsible for the disease in each family
Collect tumor specimens for histologic evaluation, culturing of intestinal organoids, and genotyping (including DNA and RNA sequencing) | End of study
  Sufficient number of tumors collected to correlate disease grade with natural history of disease and assess the variability in disease grade
Screen for occult disease and determine whether early detection affects the natural history of the disease | End of study
  Change in survival

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Wank, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caplin ME, Buscombe JR, Hilson AJ, Jones AL, Watkinson AF, Burroughs AK. Carcinoid tumour. Lancet. 1998 Sep 5;352(9130):799-805. doi: 10.1016/S0140-6736(98)02286-7. PMID 9737302
- [Background] Modlin IM, Lye KD, Kidd M. A 5-decade analysis of 13,715 carcinoid tumors. Cancer. 2003 Feb 15;97(4):934-59. doi: 10.1002/cncr.11105. PMID 12569593
- [Background] Capella C, Heitz PU, Hofler H, Solcia E, Kloppel G. Revised classification of neuroendocrine tumours of the lung, pancreas and gut. Virchows Arch. 1995;425(6):547-60. doi: 10.1007/BF00199342. PMID 7697211
- [Derived] Tang D, Lim R, Korman L, Forbes J, Ellsbury K, Auh S, Trivedi A, Chen CC, Hughes M, Wank S. Performance of capsule endoscopy for the detection of small intestinal neuroendocrine tumors in familial carcinoid: a prospective single-site study. Gastrointest Endosc. 2024 Feb;99(2):227-236. doi: 10.1016/j.gie.2023.08.024. Epub 2023 Oct 13. PMID 37838323
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-DK-0098.html